CLINICAL TRIAL: NCT07019506
Title: Evaluation of the Effectiveness of Physical Exercise on Aerobic Capacity in Patients With Cardiovascular Disease
Status: Recruiting | Type: Observational
Sponsor: Fundacion Universitaria Maria Cano (Other)
Responsible Party: Principal Investigator, Catalina Lopera Muñetón, Principal investigator MSc Clinical leadership in cancer and palliative care, Fundacion Universitaria Maria Cano
Other Study IDs: 013008002-2024-311
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Diseases; Exercise; Aerobic Capacity
Keywords: cardiovascula diseases; exercise; aerobic capacity
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cardiac rehabilitation — Sessions are conducted individually in accordance with cardiac rehabilitation guidelines, with a frequency of 2-3 times per week, each lasting 1 hour. Intensity is progressively increased on a weekly basis, with adaptations made according to each patient's specific needs. A total of 20 sessions are delivered, focused on improving the patient's cardiovascular capacity

SUMMARY:
According to the Pan American Health Organization (PAHO), non-communicable chronic diseases-primarily cardiovascular diseases-are the leading cause of death and disability worldwide. These conditions result in long-term health consequences and require significant ongoing treatment and care. Among them, ischemic heart diseases-most notably acute myocardial infarction-are highly prevalent. Globally, cardiovascular diseases are closely linked to physical inactivity as a major modifiable risk factor. In this context, exercise and physical activity have become public health priorities, with international guidelines recommending at least 150 minutes of moderate-intensity activity per week.

In Colombia, physical exercise is recognized as a key strategy for the prevention and management of non-communicable chronic diseases, as outlined in the national ten-year public health plan. However, evidence shows that few clinical services at the national or regional level consistently monitor or follow up on the proper prescription of exercise as a therapeutic strategy for cardiovascular disease management.

This study aims to describe the effectiveness of structured physical exercise on the aerobic capacity of patients with cardiovascular disease.

DETAILED DESCRIPTION:
By 2030, the United Nations Sustainable Development Goals aim to reduce premature mortality from non-communicable diseases (NCDs) by one-third. Among these, cardiovascular diseases (CVDs)-including coronary heart disease and stroke-are the most common NCDs globally.

In recent years, myocardial infarction (MI) has emerged as one of the most potentially fatal coronary events, alongside coronary artery disease (CAD). According to the World Health Organization (WHO), an estimated 17.9 million people died in 2019 from CVDs, accounting for 32% of all global deaths. Of these, approximately 85% were due to MI and stroke. In Europe, CVDs are responsible for around 4 million deaths annually, representing about 47% of total mortality, with most cases associated with coronary disease. In the United States, the American Heart Association has estimated that approximately 15 million individuals over the age of 20 live with ischemic heart disease, affecting 6.4% of the population.

In the context of cardiac rehabilitation and secondary prevention, exercise training (ET) should be a core component of rehabilitation programs for cardiac patients. Its practice has been shown to improve exercise tolerance, quality of life, functional capacity, and performance in work-related physical tasks, while also reducing cardiovascular risk factors and cardiac mortality. Several studies have demonstrated that regular physical activity significantly enhances aerobic capacity in this population, leading to reduced cardiovascular risk and improved quality of life.

In terms of metabolic equivalents (METs), improved aerobic capacity is reflected by an increased oxygen uptake during physical activity, which enables patients to perform daily tasks with less effort and reduces strain on the cardiovascular system. Moreover, adherence to exercise programs has been identified as a key factor in achieving sustainable cardiovascular health benefits. However, adherence remains a challenge, particularly among patients with chronic diseases.

For this reason, there is a need for specific exercise programs that promote the modification of risk factors, support early intervention in cardiovascular patients, and enhance adherence to therapeutic interventions. These approaches could positively impact morbidity and mortality in this population and provide critical evidence for designing more effective cardiovascular rehabilitation strategies.

Within this context, the present study aims to evaluate the effectiveness of a structured exercise program in improving the aerobic capacity of patients diagnosed with cardiovascular disease.

The benefits of therapeutic exercise (TE) on cardiac remodeling appear to occur in both early and late phases. The early remodeling phase is characterized by expansion of the infarcted area, driven by the degradation of structural collagen in the extracellular matrix (ECM) by matrix metalloproteinases (MMPs), which are secreted by immune cells in response to MI-induced inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Records between 2015 and 2024
* Men and women, between 35 and 90 years old.
* Clinical diagnosis of cardiovascular disease.
* Must be patient from Clínica el Rosario.
* Participants must have completed a baseline exercise stress test and a post-intervention stress test after the 20 sessions, and must have attended at least 90% of the prescribed sessions

Exclusion Criteria:

* Records containing incomplete data

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women, between 35 and 90 years old, residents in the metropolitan area, with a diagnosis of cardiovascular disease who entered cardiovascualr patient care program from Clínica El Rosario.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Aerobic capacity | 2015-2024
  The data will be collected from the clinical registries which have included. Aerobic capacity will be assessed through an exercise stress test, measured in metabolic equivalents (METs). Subsequently, VO₂max will be estimated using the NASA-derived formula. A poor physical fitness level will be defined as an estimated maximal oxygen consumption (VO₂max) of less than 7 METs

SECONDARY OUTCOMES:
Cardiovascular risk | 2015-2024
  The data will be collected from the clinical registries which have included Cardiovascular risk will be assessed using the American Heart Association (AHA) classification, which categorizes patients into low, moderate, high, and very high risk

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación universitaria María Cano, Medellín, Colombia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in cardiovascular diseases. Data or samples shared will be coded. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: ICF
Time Frame: Data requests can be submitted starting 12 months after article publication and the data will made accessible for up to 18 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact catalinaloperamuneton@fumc.edu.co